CLINICAL TRIAL: NCT07302581
Title: Evaluation of the Efficacy and Safety of Periodontal Ligament Integrated Implants Via Residual Periodontal Ligament Tissue in Extraction Sockets
Brief Title: Efficacy and Safety Evaluation Study of Implants With Periodontal Ligament
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OrganTech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OrgT-CPS-001; jRCTs022240055 (Registry Identifier: Japan Registry of Clinical Trials)
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Tooth Extraction; Tooth Fractures; Dental Caries; Tooth Dislocation
Keywords: Root Fracture; Crown Fracture; Tooth Mobility; Carious Tooth; Extraction site healing
MeSH Terms: conditions — Tooth Fractures; Dental Caries; Tooth Avulsion; Tooth Mobility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (1):
- Periodontal Ligament-Integrated Implant Placement (Experimental): Participants undergo preoperative evaluation, including oral examination, CT imaging, and impressions for implant simulation and fabrication. After eligibility confirmation, a single-rooted tooth is extracted using minimally invasive techniques to preserve residual periodontal ligament tissue. A periodontal ligament-integrated implant with an abutment and fixation is immediately placed into the extraction socket and stabilized with dental cement. Sutures are removed after three weeks. The implant remains unloaded for about nine weeks for healing and integration into the jawbone, with periodic radiographic evaluation. A superstructure is then fabricated and placed for controlled occlusal loading. Once integration into the jawbone via regenerated periodontal ligament is confirmed, the fixation is removed and the implant functions independently. Oral care is maintained throughout the study.
  Interventions: Device: Periodontal Ligament-Integrated Implant

INTERVENTIONS:
Device: Periodontal Ligament-Integrated Implant — The investigational device is a periodontal ligament-integrated implant designed for immediate placement into a tooth extraction socket. Unlike conventional osseointegrated implants, this device utilizes residual periodontal ligament tissue to establish functional attachment and physiological integration with the alveolar bone. The implant-abutment assembly is stabilized with a temporary fixation device for approximately nine weeks, during which integration into the jawbone through the residual periodontal ligament is promoted. After the healing phase, a definitive superstructure is fabricated and placed to allow controlled occlusal loading. Once integration into the jawbone and implant stability are confirmed, the fixation device is removed, and the implant functions independently. The device remains unapproved and is evaluated for safety and efficacy in this study.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of periodontal ligament-integrated implants placed via residual periodontal ligament tissue in extraction sockets in adult patients (aged 18 and older) requiring extraction of a single-rooted tooth.

The main questions it aims to answer are:

* Does the periodontal ligament-integrated implant achieve stable integration with the jawbone at 24 weeks after placement?
* Can this implant reproduce physiological tooth mobility and sensory function similar to natural teeth while maintaining periodontal health?

This is a multicenter, single-arm, exploratory study with approximately six participants.

Participants will:

* Undergo tooth extraction of one single-rooted tooth that meets eligibility criteria.
* Receive immediate placement of a periodontal ligament-integrated implant into the extraction socket.
* Attend scheduled follow-up visits over 48 weeks for assessments including:

  * Dental X-rays and clinical examinations to evaluate bone healing, periodontal ligament formation, and implant stability.
  * Measurements of tooth mobility, pocket depth, and pain levels.
  * Quality of life assessments using a standardized oral health questionnaire.

Researchers will monitor participants for implant integration, safety outcomes, and physiological function restoration over the study period.

DETAILED DESCRIPTION:
This multicenter, single-arm exploratory clinical trial investigates the efficacy and safety of periodontal ligament (PDL)-integrated implants placed immediately after tooth extraction, using residual periodontal ligament tissue within the extraction socket to achieve functional attachment. The investigational device is an unapproved medical implant designed to reproduce physiological tooth function by utilizing the periodontal tissue for anchorage and sensory integration, unlike conventional osseointegrated implants that rely solely on bone integration.

The rationale for this study is that preserving and integrating residual PDL tissue may allow the implant to develop a PDL-like attachment, potentially restoring physiological tooth mobility, mechanosensory feedback, and natural load distribution to the alveolar bone. This could enable improved long-term function and compatibility with adjacent natural teeth, particularly in cases where the implant is connected to them.

Participants will undergo immediate implant placement following extraction of a single-rooted tooth (incisor to premolar) that meets inclusion criteria. The implant-abutment assembly is secured temporarily using a fixation device to ensure stability during early healing. The fixation is maintained for approximately 9 weeks, followed by staged removal and functional loading through placement of a superstructure. Throughout the observation period (up to 48 weeks), multiple evaluations will be conducted to assess integration into the jawbone, periodontal attachment formation, bone remodeling, implant mobility, and patient-reported comfort.

Comprehensive radiographic, clinical, and physiological assessments will be performed to monitor healing dynamics, bone response, and periodontal adaptation. Safety will be assessed by recording adverse events related to surgery, device performance, or oral function. Oral hygiene and supportive care will be provided throughout the study.

The findings from this exploratory research are expected to provide foundational data regarding the biological feasibility, mechanical behavior, and clinical safety of PDL-integrated implants as a novel approach for immediate implant placement and restoration of physiological dental function.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have only one single-rooted tooth, from the upper or lower incisors to the premolars, which require extraction due to caries or a fracture, and who have healthy periodontal tissue remaining around the root of the tooth to be extracted.
* The teeth adjacent to the tooth to be extracted are natural teeth with healthy periodontal tissues, and no abnormalities are found in dental X-rays, CT scans, periodontal pocket examinations, or physiological mobility tests. Also, patients should be able to achieve proper occlusion with opposing teeth.
* Patients aged 18 years or older at the time of consent.
* Patients who have provided written consent to participate in this clinical study and are able to comply with study visits and procedures.

Exclusion Criteria:

* Patients whose jawbone is still growing.
* Patients undergoing orthodontic treatment or wearing retainers after orthodontic treatment.
* Patients with multiple missing teeth or an edentulous jaw where multiple occlusal support areas of the remaining teeth are missing.
* Patients who have periodontal pockets of 4mm or more around the root of the tooth to be extracted or the teeth adjacent to the tooth to be extracted.
* Patients with bacterial infection or acute inflammation such as periodontitis in the tooth to be extracted.
* Patients with apical periodontitis in the tooth to be extracted.
* Patients who will have two or more consecutive missing teeth or free-end edentulous space due to the extraction of the target teeth.
* Patients who have already had the target tooth extracted.
* Patients for whom extraction of the target tooth is expected to be difficult.
* Patients who are not healthy enough to undergo the tooth extractions and surgical procedures required for implant treatment using this product.
* Patients with abnormal root morphology or position (curved, tilted, etc.) of the tooth to be extracted.
* Patients in whom this product cannot be implanted due to the root size of the tooth to be extracted (root length less than 10 mm, root diameter at the cervical part less than 5.4 mm in long diameter, less than 3.4 mm in short diameter) or malocclusion.
* Patients with open bite.
* Patients with a history of hypersensitivity to the components of this product or similar products.
* Patients with alveolar bone resorption in the area where the implant is to be placed.
* Patients with bleeding disorders. (There is a risk of abnormal bleeding and poor healing of the surgical site).
* Patients with uncontrolled diabetes. (There is a risk of poor healing of the surgical site and increased susceptibility to infection.)
* Patients for whom general oral surgery is contraindicated. (There is a risk that the invasive procedure may worsen the disease, cause recurrence of preexisting conditions, or result in poor healing of the surgical site postoperatively.)
* Patients who undergo radiation therapy or chemotherapy due to malignant tumors, etc. (There is a risk that the surgical site may not heal properly.)
* Patients receiving bisphosphonate therapy.
* Patients who currently smoke.
* Patients who do not understand or cooperate with the treatment.
* Pregnant patients or patients who may be pregnant.
* Any other patient deemed unsuitable for participation in this study by the principal investigator (or co-investigator).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Rate of integration into the jawbone at 24 Weeks Post-Implantation | 24 weeks after implantation
  Presence or absence of integration with the jawbone at 24 weeks postoperatively (Rate of integration into the jawbone).

SECONDARY OUTCOMES:
Rate of integration into the jawbone Over Time | 9, 18, and 48 weeks postoperatively
  Presence or absence of integration into the jawbone (9 weeks postoperatively, 18 weeks postoperatively, 48 weeks postoperatively).
Periodontal Pocket Depth | Baseline (approximately 11 weeks preoperative) to 48 weeks postoperatively
  Periodontal pocket depth (mm) at Baseline (Visit 1 - approximatelly 11 weeks preoperative), and at 9, 18, 24, and 48 weeks postoperatively.
Physiological Instability (PT value) With Fixation | Immediately after surgery to 36 weeks postoperatively
  Physiological instability (periotest value) immediately after surgery, 1 week after surgery, 3 weeks after surgery, 7 weeks after surgery, 9 weeks after surgery, 10 weeks after surgery, 14 weeks after surgery, 18 weeks after surgery, 24 weeks after surgery, and 36 weeks after surgery with fixation.
Physiological Tooth Mobility (PT Value) Without Fixation | Baseline (approximately 11 weeks preoperative) to 48 weeks postoperatively
  Physiological tooth mobility (periotest value) without fixation, measured at Baseline (approximately 11 weeks preoperatively) (Visit 3), and at 9, 18, 24, 36, and 48 weeks postoperatively, as well as clinical tooth mobility (Miller classification) assessed by the surgeon.
Perceptual and Sensory Evaluation (Pain) | Baseline (approximately 11 weeks preoperatively) to 48 weeks postoperatively
  Perceptual and sensory evaluation (pain) using the numerical rating scale, conducted at Baseline (approximately 11 weeks preoperatively) (Visit 3), the day after surgery, and at 1, 3, 7, 9, 10, 14, 18, 24, 36, and 48 weeks postoperatively.
Peri-Implant Bone Augmentation and Vertical Bone Resorption | Baseline (approximately 11 weeks preoperatively) to 48 weeks postoperatively
  Peri-implant bone augmentation (formation) and vertical bone resorption (dental X-ray) assessed at Baseline (approximately 11 weeks preoperatively) (Visit 1), immediately after surgery, and at 3, 7, 9, 14, 18, 24, and 48 weeks postoperatively.
Formation of Periodontal Ligament Space | 7 to 48 weeks postoperatively
  Formation of the periodontal ligament space around the implant (dental X-ray), assessed at 7, 9, 14, 18, 24, and 48 weeks postoperatively.

OTHER OUTCOMES:
Oral Related QOL (Japan Prosthodontic Society Questionnaire) | Baseline (approximately 11 weeks preoperatively) to 48 weeks postoperatively
  Oral related QOL (Japan Prosthodontic Society questionnaire), assessed at Baseline (approximately 11 weeks preoperatively) (Visit 3), and at 18 and 48 weeks postoperatively.
Safety Evaluation - Incidence of adverse events and device-related defects | From implantation to 48 weeks postoperatively
  Incidence of diseases and frequency of defects.

CONTACTS AND LOCATIONS:
Overall Officials: Shohei Kasugai, PhD, Study Director — Minami Tohoku Medical Clinic
Locations (2):
- Japan (2):
  - Minami Tohoku Medical Clinic, Kōriyama, Fukushima
  - Hillside Akasaka Dental Clinic, Minato-Ku, Tokyo

IPD SHARING:
Plan to Share IPD: No